CLINICAL TRIAL: NCT00207389
Title: A Pilot Study to Examine the Relationship Between Changes in Plasma GIP Levels and Other Gastrointestinal Peptides Following Gastric Bypass Surgery in Obese Patients
Brief Title: A Study to Examine Changes in GIP Plasma Levels Following Gastric Bypass Surgery in Obese Patients
Status: Terminated | Type: Observational
Why Stopped: Insufficient funding
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Caroline Apovian, Principal Investigator, Boston Medical Center
Other Study IDs: H-22610
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Type 2 Diabetes Mellitus; Insulin Resistance
Keywords: Incretins:GIP , GLP-1; Gastric bypass surgery; Laparoscopic gastric bypass surgery; Postprandial expression of GIP
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic gastric bypass: Patients undergoing Laparoscopic gastric bypass
- Open gastric bypass: Patients undergoing Open gastric bypass

SUMMARY:
Obesity is a multinational epidemic. There is evidence that despite educational measures and increased public awareness, the number of obese individuals continues to increase. Of the numerous obesity-related comorbidities, type 2 diabetes remains one of the most significant in terms of mortality and health care costs. Gastric Bypass Surgery (GBS) not only offers an effective form of therapy for morbid obesity, but also amelioration of type 2 diabetes mellitus. The normalization of glucose levels in GBS patients occurs within days after surgery and has been shown in surgical literature to be independent of the weight loss after surgery. The proximal gut, the site of release of certain incretins, may play a role in glucose homeostasis in obese individuals with type 2 diabetes mellitus. One such incretin is GIP, which when released into the circulation during the immediate postprandial period, accentuates the insulin response to a glucose meal. It is hypothesized that overactivity of this enteroinsular axis in obese individuals produces cell resistance to insulin and subsequent type 2 diabetes mellitus. A previous study reported elevated fasting GIP levels, as well as an exaggerated GIP response to a glucose meal, in obese subjects, which was significantly reduced months after GBS following weight loss. This pilot study of obese patients scheduled for GBS will compare the serum levels of certain peptides, including GIP, following a glucose meal before and after GBS, before weight loss has occured. In order to reproduce the preoperative state, and therefore to demonstrate the physiologic change, a small group of subjects who undergo open surgery will undergo the same measurements after surgery, but using a model in which the meal traverses the stomach, duodenum and jejunum with the aid of a gastrostomy tube.

DETAILED DESCRIPTION:
This is a pilot study to collect the relevant information for planning a larger and more definitive investigation. A total of thirty subjects will be evaluated in this study to be conducted at the Boston Medical Center. The study population will consist of obese patients who meet the criteria and have been scheduled by their surgeon for GBS. We plan to enroll a total of 30 subjects scheduled for GBS. Patients will be assigned according to standard surgical care to either open or laparoscopic surgery. We plan to enroll 20 subjects who undergo laparoscopic GBS (LAP) and 10 subjects who undergo open GBS (OPEN). All potential subjects will have undergone baseline screening as a part of their routine medical evaluation performed by Dr. Apovian or Dr. McDonnell in the Nutrition Center at BMC. This standard testing includes medical history, physical examination, complete blood count, serum electrolytes, BUN, creatinine, fasting blood glucose and glycosylated hemoglobin. If patients are identified as having type 2 diabetes or glucose intolerance, they will be provided informed consent. If consented subjects meet all the inclusion and exclusion criteria, each will undergo a baseline oral glucose tolerance test (OGTT) approximately one week before surgery. Plasma concentrations of insulin, GIP, glucagon, and GLP-1 will also be measured along with glucose levels and other peptides (CCK, ghrelin, c-peptide) at the same intervals, using commercially available assay kits. Post-operatively, subjects in the LAP group will undergo 2 OGTTs, while subjects in the OPEN group will undergo 2 OGTTs and one glucose tolerance test through the gastrostomy tube (GGTT). The results of the postoperative OGTTs will be compared with baseline OGTTs. In a separate analysis, the results of the GGTTs will be compared with the baseline and postoperative OGTTs.

Inclusion criteria Patients 21-64 y ears of age with obesity (defined as a body mass index, BMI, > or = 30) and type 2 diabetes or impaired glucose tolerance, who have been selected and scheduled for gastric bypass surgery.

Exclusion criteria Substance abuse, consumption of more than two alcoholic drinks per day, use of more than 20 units of insulin (any brand or type) per day, and having a fasting blood glucose >180mg/dl on screening bloodwork.

F2. Procedure

All subjects will undergo a total of 3 OGTTs, 1 before surgery and 2 after. The OPEN group will also have a glucose tolerance test via a gastrostomy tube (GGTT) placed in the duodenum (per routine surgical procedure) as described below. The OGTT consists of a 12-hour overnight fast followed by drinking a 225 ml of solution containing 75 grams of a glucose (Glucola), over 30 minutes. 30 minutes is the average time a patient requires in order to drink a 225ml Glucola drink after gastric bypass surgery. In order to be able to make a valid comparison of the three OGTTs, each OGTT will require that the subject drink over 30 minutes. Blood samples are obtained from an intravenous catheter at various time intervals: 5 minutes and immediately before drinking the Glucola, and 5, 10, 15, 30, 60, 90, 120, and 180 minutes afterwards. Blood levels of glucose, insulin, glucose-dependent insulinotropic polypeptide (GIP), glucagon, and Glucagon-Like Peptide (GLP-1), CCK, ghrelin and c-peptide will be determined from the samples obtained. In addition, at hour 2 during the OGTT (when glucose peaks) we will obtain a real-time glucose level with a drop of blood from the indwelling line. The GGTT follows that same protocol as the OGTT, but the Glucola is administered via a gastrostomy tube, placed per routine surgical procedure in patients undergoing open GBS. Approximately 1 week before surgery, all subjects will undergo an OGTT in the GCRC. Between day 6 and 10 after their surgery, when subjects are tolerating their standard 240cc liquid meals 3-4 times daily, subjects will undergo the third OGTT. Although most subjects are discharged on day 3 or 4 after surgery, and will be asked to return to the GCRC, those subjects who remain in the hospital through day 5 will have the option to remain in the hospital for an additional time (1-2 days) or to go home and return to the GCRC within 5 days (no later than POD 10) The additional hospital days will be paid for by the GCRC. After surgery, subjects in LAP group will have one OGTT. Subjects in the OPEN group will have a GGTT on one day and an OGTT on the following day. Subjects will be weighed before surgery and every day during the first week after surgery and before each glucose tolerance test. All subjects will undergo a final OGTT approximately 3 -4 weeks after surgery. This will take place in the GCRC on the same day as a routine follow up visit to their surgeon.

Patients will be contacted by telephone for assessment approximately 24 hours before and after each GTT.

There are 2 primary outcomes: 1) Change in plasma GIP response to glucose after GBS and 2) change in insulin sensitivity after GBS, as measured by an area-under-the-curve equation for a standardized 180-minute oral glucose tolerance test. Secondary outcomes include 1) Change in plasma GLP-1 response to glucose after GBS and 2) change in plasma glucagon response to glucose after GBS, as measured by the equation used for the primary outcome.

We expect that our enrollment period will be 18 months to 24 months. The estimated duration of the entire study is 28 months

ELIGIBILITY:
Inclusion Criteria:

* Patients 21-64 years of age
* Obese (defined as a body mass index, BMI, > or = 30)
* Type 2 diabetes or impaired glucose tolerance
* Have been selected and scheduled for gastric bypass surgery.

Exclusion Criteria:

* Substance abuse
* Consumption of more than two alcoholic drinks per day
* Use of more than 20 units of insulin (any brand or type) per day
* Fasting blood glucose >180mg/dl on screening bloodwork.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2004-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
GIP area under the curve after OGTT

SECONDARY OUTCOMES:
Other GI peptides and hormones after OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Apovian, MD, Principal Investigator — Boston University Medical Cneter; Michael Wolfe, MD, Principal Investigator — Boston University; Marie Mcdonnell, MD, Study Chair — Boston University; Harmony Allison, MD, Study Chair — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] MCINTYRE N, HOLDSWORTH CD, TURNER DS. NEW INTERPRETATION OF ORAL GLUCOSE TOLERANCE. Lancet. 1964 Jul 4;2(7349):20-1. doi: 10.1016/s0140-6736(64)90011-x. No abstract available. PMID 14149200
- [Background] Miyawaki K, Yamada Y, Ban N, Ihara Y, Tsukiyama K, Zhou H, Fujimoto S, Oku A, Tsuda K, Toyokuni S, Hiai H, Mizunoya W, Fushiki T, Holst JJ, Makino M, Tashita A, Kobara Y, Tsubamoto Y, Jinnouchi T, Jomori T, Seino Y. Inhibition of gastric inhibitory polypeptide signaling prevents obesity. Nat Med. 2002 Jul;8(7):738-42. doi: 10.1038/nm727. Epub 2002 Jun 17. PMID 12068290
- [Background] Bayliss WM, Starling EH. Croonian lecture. The chemical regulation of the secretory process. Proc R Soc Lond 1904(73):310-332.
- [Background] GREGORY RA, TRACY HJ. THE CONSTITUTION AND PROPERTIES OF TWO GASTRINS EXTRACTED FROM HOG ANTRAL MUCOSA. Gut. 1964 Apr;5(2):103-14. No abstract available. PMID 14159395
- [Background] Jorpes E, Mutt V. Cholecystokinin and pancreozymin, one single hormone? Acta Physiol Scand. 1966 Jan-Feb;66(1):196-202. doi: 10.1111/j.1748-1716.1966.tb03185.x. No abstract available. PMID 5935672
- [Background] Kosaka T, Lim RKS. Demonstration of the humoral agent in fat inhibited gastric secretion. Proc Soc Exp Biol Med 1930;27:890-891.
- [Background] Brown JC, Pederson RA, Jorpes E, Mutt V. Preparation of highly active enterogastrone. Can J Physiol Pharmacol. 1969 Jan;47(1):113-4. doi: 10.1139/y69-020. No abstract available. PMID 5761841
- [Background] Cleator IG, Gourlay RH. Release of immunoreactive gastric inhibitory polypeptide (IR-GIP) by oral ingestion of food substances. Am J Surg. 1975 Aug;130(2):128-35. doi: 10.1016/0002-9610(75)90360-8. No abstract available. PMID 1098505
- [Background] Villar HV, Fender HR, Rayford PL, Bloom SR, Ramus NI, Thompson JC. Suppression of gastrin release and gastric secretion by gastric inhibitory polypeptide (GIP) and vasoactive intestinal polypeptide (VIP). Ann Surg. 1976 Jul;184(1):97-102. doi: 10.1097/00000658-197607000-00016. PMID 938120
- [Background] Arnold R, Creutzfeldt W, Ebert R, Becker HD, Borger HW, Schafmayer A. Serum gastric inhibitory polypeptide (GIP) in duodenal ulcer disease: relationship to glucose tolerance, insulin, and gastrin release. Scand J Gastroenterol. 1978;13(1):41-7. doi: 10.3109/00365527809179804. PMID 635445